CLINICAL TRIAL: NCT00448526
Title: Effect of Low Protein Diet in Preventing the Progression of Diabetic Nephropathy
Acronym: LPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated: recruiting or enrolling participants has halted and will not resume because low protein diet is not feasible nor efficious.
Sponsor: Kanazawa Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H8-H-077
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Diabetic Nephropathies
Keywords: Low protein diet, type 2 Diabetic nephropathy; Comparing the effect of Low protein Diet on diabetic nephropathy to that of normal protein diet
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: low protein diet

SUMMARY:
Diabetic nephropathy is the leading cause of chronic kidney disease all the world in spite of progress in new treatment for diabetes and anti hypertensive drugs. Additional treatments are thus needed to arrest the progression of diabetic nephropathy. Although there is insufficient evidence to suggest that a low-protein diet improves renal dysfunction, it is recommended as a mainstay of nutritional management. We here assessed the role of low protein diet in renal function as well as albuminuria in type 2 diabetic patients with nephropathy for a median of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Urinary protein excretion 1-10 g/day
* Serum Cr <2.0 mg/dl
* With diabetic retinopathy > SDR
* Normal protein intake instruction
* Patients whose consent is obtained at >20 or age =<65

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Non-diabetic nephropathy
* Urinary tract infection
* Congestive heart failure
* Unstable angina
* Myocardial infarction
* Stroke
* Severe hepatopathy
* Life threatening disease such as malignant tumor
* Patients on ACE-I and or ARB treatment
* Patients on instruction of low protein diet
* BW< 80% of IBW
* Pregnant, lactating, and probably pregnant patients
* Patients judged as being inappropriate fir the subjects

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1997-12; Study Completion 2006-08

PRIMARY OUTCOMES:
annual change of GFR
annual change of Ccr
annual change of 1/Cr
incidence rate of the doubling of sCr
time to the doubling of sCr

SECONDARY OUTCOMES:
urinary albumin and protein excretion
% change of urinary albumin and protein excretion from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ryuichi Kikkawa, M.D., Study Director — Shiga University of Medical Science

REFERENCES:
- [Derived] Jiang S, Fang J, Li W. Protein restriction for diabetic kidney disease. Cochrane Database Syst Rev. 2023 Jan 3;1(1):CD014906. doi: 10.1002/14651858.CD014906.pub2. PMID 36594428
- [Derived] Koya D, Haneda M, Inomata S, Suzuki Y, Suzuki D, Makino H, Shikata K, Murakami Y, Tomino Y, Yamada K, Araki SI, Kashiwagi A, Kikkawa R; Low-Protein Diet Study Group. Long-term effect of modification of dietary protein intake on the progression of diabetic nephropathy: a randomised controlled trial. Diabetologia. 2009 Oct;52(10):2037-45. doi: 10.1007/s00125-009-1467-8. Epub 2009 Aug 4. PMID 19652945